CLINICAL TRIAL: NCT02581631
Title: A Phase I/ II Study to Evaluate the Safety and Preliminary Efficacy of Nivolumab in Combination With Brentuximab Vedotin in Subjects With Relapsed Refractory Non Hodgkin Lymphomas With CD30 Expression (CheckMate 436: CHECKpoint Pathway and Nivolumab Clinical Trial Evaluation 436)
Brief Title: An Investigational Immuno-therapy Safety and Effectiveness Study of Nivolumab in Combination With Brentuximab Vedotin to Treat Non-Hodgkin Lymphomas
Acronym: CheckMate 436
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-436; 2015-003286-28 (EudraCT Number)
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Non-Hodgkin's Disease
MeSH Terms: interventions — Nivolumab; Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab+Brentuximab Vedotin (Experimental): Nivolumab+Brentuximab Vedotin dose as specified
  Interventions: Biological: Nivolumab; Drug: Brentuximab Vedotin

INTERVENTIONS:
Biological: Nivolumab
Drug: Brentuximab Vedotin

SUMMARY:
The purpose of this study is to determine whether Nivolumab, in combination with brentuximab vedotin, is safe and effective in patients with certain subtypes of non-Hodgkin's lymphomas with CD30 expression that have not responded to treatment or have come back. The subtypes we are studying are Diffuse Large B-Cell Lymphoma (DLBCL), Peripheral T-Cell Lymphoma (PTCL), Cutaneous T-Cell Lymphoma (CTCL), Primary Mediastinal Large B-Cell Lymphoma (PMBL) and Mediastinal Gray Zone Lymphoma (MGZL).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Relapsed/refractory diffuse large B cell lymphoma (DLBCL), relapsed/refractory peripheral T cell lymphoma (PTCL) (all subtypes excluding anaplastic large cell lymphoma), relapsed/refractory Cutaneous T cell lymphoma (CTCL) mycosis fungoides/sezary syndrome (MF/SS), relapsed/refractory primary mediastinal B lymphoma (PMBL), and relapsed/refractory mediastinal gray zone lymphoma (MGZL)
* Expression of CD30
* Subjects must be 18 years or older (≥ 15 years for PMBL)

Exclusion Criteria:

* Known central nervous system (CNS) lymphomas; Active cerebral/meningeal disease related to the underlying malignancy
* Active, known, or suspected autoimmune disease

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-02-11 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (16):
  - Local Institution - 0017, Birmingham, Alabama
  - University Of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Local Institution - 0012, Tampa, Florida
  - Winship Cancer Institute., Atlanta, Georgia
  - University Of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - Local Institution - 0003, New York, New York
  - Local Institution - 0010, New York, New York
  - University Of Rochester, Rochester, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Portland Medical Center, Portland, Oregon
  - Bon Secours-St Francis Hosp, Greenville, South Carolina
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (3):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Local Institution - 0011, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- France (2):
  - Hopital Saint Louis, Paris
  - Local Institution - 0020, Pierre-Bénite
- Italy (3):
  - Local Institution - 0018, Bergamo
  - Local Institution - 0024, Bologna
  - Istituto Clinico Humanitas, Rozzano (milano)
- Local Institution - 0027, Hospitalet de Llobregat - Barcelona, Spain
- United Kingdom (2):
  - Churchill Hospital, Oxford, Oxfordshire
  - Royal Marsden Hospital, Sutton, Surrey

REFERENCES:
- [Derived] Zinzani PL, Santoro A, Gritti G, Brice P, Barr PM, Kuruvilla J, Cunningham D, Kline J, Johnson NA, Mehta-Shah N, Lisano J, Wen R, Akyol A, Moskowitz AJ. Nivolumab combined with brentuximab vedotin for R/R primary mediastinal large B-cell lymphoma: a 3-year follow-up. Blood Adv. 2023 Sep 26;7(18):5272-5280. doi: 10.1182/bloodadvances.2023010254. PMID 37352266
- [Derived] Zinzani PL, Santoro A, Gritti G, Brice P, Barr PM, Kuruvilla J, Cunningham D, Kline J, Johnson NA, Mehta-Shah N, Manley T, Francis S, Sharma M, Moskowitz AJ. Nivolumab Combined With Brentuximab Vedotin for Relapsed/Refractory Primary Mediastinal Large B-Cell Lymphoma: Efficacy and Safety From the Phase II CheckMate 436 Study. J Clin Oncol. 2019 Nov 20;37(33):3081-3089. doi: 10.1200/JCO.19.01492. Epub 2019 Aug 9. PMID 31398081
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Dose Evaluation Phase (Cohort A) will include a dose limiting toxicity (DLT) evaluation for the dose level of brentuximab vedotin 1.8 mg/kg in combination with nivolumab 240 mg. The reduced dose of brentuximab vedotin at 1.2 mg/kg was not needed based on the safety data reviewed throughout the DLT evaluation period.
Groups:
- Diffuse Large B-cell Lymphoma (DLBCL); Peripheral T-cell Lymphoma (PTCL); Cutaneous T-cell Lymphoma (CTCL); Mediastinal Grey Zone Lymphoma (MGZL); Primary Mediastinal B-cell Lymphoma (PMBL): 1.8mg/kg brentuximab vedotin (BV) + 240mg nivolumab
Period: Overall Study
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Started | 42 | 33 | 29 | 10 | 30
Phase 1 DLT Evaluable Participants | 2 | 1 | 3 | 0 | 0
Completed Phase 1 DLT Evaluation | 2 | 1 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 42 | 33 | 29 | 10 | 30
Not completed — Disease progression | 29 | 19 | 13 | 5 | 8
Not completed — Study drug toxicity | 4 | 6 | 7 | 0 | 3
Not completed — AE unrelated to study drug | 3 | 1 | 1 | 0 | 2
Not completed — Request to discontinue | 1 | 0 | 3 | 0 | 1
Not completed — participant withdrew consent | 3 | 0 | 1 | 0 | 0
Not completed — Maximum clinical benefit | 1 | 7 | 1 | 3 | 13
Not completed — Other Reasons | 1 | 0 | 2 | 2 | 3
Not completed — Poor/Non-Compliance | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL) | Total
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (13.2) | 59.1 (12.0) | 57.9 (12.39) | 39.9 (15.2) | 37.3 (12.9) | 52.6 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 11 | 13 | 4 | 17 | 65
  Male | 22 | 22 | 16 | 6 | 13 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 0 | 1 | 4
  Not Hispanic or Latino | 14 | 13 | 16 | 6 | 9 | 58
  Unknown or Not Reported | 27 | 18 | 13 | 4 | 20 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 5 | 1 | 2 | 13
  White | 36 | 30 | 24 | 9 | 26 | 125
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety Analysis - Number of Participants With Dose Limiting Toxicities (DLT) in the DLT Evaluation Phase
Description: DLTs are defined as any study drug-related toxicity (brentuximab vedotin or nivolumab) that requires either a dose reduction or delay of more than 7 days of either study drug in Cycle 2 or delays the Cycle 3 Day 1 administration of combined treatment by more than 7 days.
Time Frame: From first dose of treatment to 6 weeks after first dose
Population: DLT evaluable Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 2 | 1 | 3 | 0 | 0
Participants | 0 | 0 | 0 |  |

2. Primary Outcome: Safety Analysis - Number of Participant Deaths
Description: Number of participant Deaths
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in Cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 24 | 22 | 3 | 3 | 5

3. Primary Outcome: Safety Analysis - Number of Participants With Adverse Advents
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 42 | 33 | 29 | 10 | 30

4. Primary Outcome: Safety Analysis - Number of Participants With Serious Adverse Events
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * results in death
  * is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * requires inpatient hospitalization or causes prolongation of existing hospitalization.
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 22 | 19 | 14 | 4 | 10

5. Primary Outcome: Safety Analysis - Number of Participants With Adverse Events Leading to Discontinuation
Description: Number of participants with adverse events leading to discontinuation
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 11 | 10 | 6 | 2 | 8

6. Primary Outcome: Safety Analysis - Number of Participants With Adverse Events Leading to Dose Delay or Reduction
Description: Number of participants with adverse events leading to dose delay or reduction
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 16 | 15 | 14 | 3 | 17

7. Primary Outcome: Safety Analysis - Number of Participants With Drug Related Adverse Events
Description: Number of participants with Drug Related Adverse Events
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants in cohort B
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 35 | 27 | 25 | 9 | 25

8. Primary Outcome: Safety Analysis - Percentage of Participants With Thyroid Test Abnormalities
Description: Percentage of participants with specific thyroid test abnormalities
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants with at least one on treatment TSH measurement
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 26 | 27 | 22 | 9 | 25
Percentage of Participants
  TSH > ULN | 34.6 | 29.6 | 18.2 | 11.1 | 24.0
  TSH > ULN w/ TSH ≤ ULN at baseline | 26.9 | 22.2 | 18.2 | 0 | 8.0
  TSH > ULN w/at least 1 FT3/FT4 value < LLN | 11.5 | 11.1 | 13.6 | 0 | 4.0
  TSH > ULN w/all other FT3/FT4 values ≥ LLN | 15.4 | 11.1 | 0 | 11.1 | 8.0
  TSH > ULN with FT3/FT4 testing missing | 7.7 | 7.4 | 4.5 | 0 | 12.0
  TSH < LLN | 7.7 | 7.4 | 4.5 | 11.1 | 24.0
  TSH < LLN w/TSH ≥ LLN at baseline | 7.7 | 0 | 4.5 | 0 | 20.0
  TSH < LLN w/at least 1 FT3/FT4 value > ULN | 0 | 3.7 | 4.5 | 0 | 20.0
  TSH < LLN w/ all other FT3/FT4 values ≤ ULN | 0 | 3.7 | 0 | 11.1 | 0
  TSH < LLN w/ FT3/FT4 test missing | 7.7 | 0 | 0 | 0 | 4.0

9. Primary Outcome: Safety Analysis - Percentage of Participants With Liver Test Abnormalities
Description: Percentage of participants with specific Liver test abnormalities
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Percentage of Participants
  ALT or AST > 3 x ULN | 4.8 | 6.1 | 13.8 | 20.0 | 24.0
  ALT or AST > 5 x ULN | 2.4 | 0 | 6.9 | 10.0 | 10.0
  ALT or AST > 10 x ULN | 0 | 0 | 0 | 10.0 | 6.7
  ALT or AST > 20 x ULN | 0 | 0 | 0 | 10.0 | 6.7
  Total Bilirubin > 2 x ULN | 0 | 6.1 | 3.4 | 20.0 | 3.3
  ALT or AST elevation > 3 x ULN w/Bilirubin > 2 x ULN within 1 day | 0 | 3.0 | 3.4 | 10.0 | 3.3
  ALT or AST elevation > 3 x ULN w/Bilirubin 2 x ULN within 30 days | 0 | 3.0 | 3.4 | 10.0 | 3.3

10. Primary Outcome: Objective Response Rate (ORR)
Description: The percentage of participants with a best overall response (BOR) of CR or PR.
  DLBCL, PTCL, PMBL & MGZL complete and partial response are outlined in the Lugano Classification 2014 and Lymphoma Response to Immunomodulatory therapy Criteria.
  CTCL complete and partial response are defined in The consensus Global Response Score assessment.
Time Frame: CTCL: 20 Months, PTCL: 26.5 Months, DLBCL: 26 Months, MGZL: 30 Months and PMBL 25.5 Months
Population: All Treated Participants
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Percentage of participants | 28.6 [19.4 to 39.4] | 45.5 [33.3 to 58.0] | 41.4 [28.8 to 55.0] | 70.0 [44.8 to 88.4] | 73.3 [60.3 to 83.8]

11. Secondary Outcome: Duration of Response (DOR)
Description: DOR will be calculated from the date of initial documentation of a response (CR, or PR) to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death due to any cause, whichever occurs first.
  DLBCL, PTCL, PMBL & MGZL complete and partial response are outlined in the Lugano Classification 2014 and Lymphoma Response to Immunomodulatory therapy Criteria.
  CTCL complete and partial response are defined in The consensus Global Response Score assessment.
Time Frame: From the first patient first visit to 8 months after the last patient first visit (up to 48 months)
Population: All Treated Participants who achieve a partial response or complete response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 12 | 15 | 12 | 7 | 22
Months | 3.55 [1.18 to 36.53] | 4.60 [2.76 to 12.75] | 26.97 [2.79 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, the upper limit number is simply undefined, and denoted as NA. | 20.76 [1.22 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, the upper limit number is simply undefined, and denoted as NA. | NA [23.33 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, then median DOR and upper limit number is simply undefined, and denoted as NA.

12. Secondary Outcome: Complete Response Rate (CRR)
Description: The CRR is defined as the percentage of participants with a BOR (Best overall response) of CR divided by the number of treated participants.
  DLBCL, PTCL, PMBL & MGZL (CR)
  1.Complete disappearance of all detectable clinical evidence of disease. 2.Bone marrow: No evidence of FDG- avid disease in marrow. CTCL (CR)
  1. 100% clearance of skin lesions.
  2. all lymph nodes ≤1.5 cm, N3 classification and ≤ 1.5 cm in their long axis and > 1 cm in their short axis at baseline, must be ≤ 1 cm in their short axis or biopsy negative for lymphoma.
  3. organs should not be enlarged on examination or imaging
  4. absence of blood involvement
Time Frame: From first dose to the date of initial objectively documented progression or the date of subsequent therapy, whichever occurs first (up to 48 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Percentage of Participants | 7.1 | 33.3 | 3.4 | 50.0 | 40.0

13. Secondary Outcome: Duration of Complete Response
Description: The duration of CR will only be evaluated in participants with BOR of CR and is defined as the time from first documentation of CR to the date of relapse or death due to any cause, whichever occurs first.
  DLBCL, PTCL, PMBL & MGZL (CR)
  1.Complete disappearance of all detectable clinical evidence of disease. 2.Bone marrow: No evidence of FDG- avid disease in marrow. CTCL (CR)
  1. 100% clearance of skin lesions.
  2. all lymph nodes ≤1.5 cm, N3 classification and ≤ 1.5 cm in their long axis and > 1 cm in their short axis at baseline, must be ≤ 1 cm in their short axis or biopsy negative for lymphoma.
  3. organs should not be enlarged on examination or imaging
  4. absence of blood involvement
Time Frame: From first dose to the date of relapse or death due to any cause, whichever occurs first. (about 48 months)
Population: All Treated Participants who achieved a complete response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 3 | 11 | 1 | 5 | 12
Months | 36.53 [9.92 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, upper limit number is simply undefined, and denoted as NA. | 7.39 [2.17 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, upper limit number is simply undefined, and denoted as NA. | NA [NA to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, then median DOR and upper limit number is simply undefined, and denoted as NA. | NA [NA to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, then median DOR, lower limit number and upper limit number is simply undefined, and denoted as NA. | NA [27.89 to NA] — The median DOR is defined to be the time at which 50% of treated participants achieved a response. If the number of responders doesn't reach 50% at the end of the available data, then median DOR and upper limit number is simply undefined, and denoted as NA.

14. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death due to any cause, whichever comes first. Participants who are progression-free and alive or have unknown status will be censored at the last tumor assessment. Participants who did not have any onstudy tumor assessments and did not die will be censored on the date of first treatment. For participants who received subsequent therapy prior to documented progression, it will be censored on the last tumor assessment date prior to or on subsequent therapy.
Time Frame: From first dose of study drug until the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death due to any cause, whichever comes first. (about 48 months)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Months | 2.60 [1.38 to 2.79] | 4.30 [1.58 to 5.62] | 15.61 [4.86 to NA] — Insufficient number of events to calculate using the K-M method | 21.88 [0.07 to NA] — Insufficient number of events to calculate using the K-M method | 25.95 [2.63 to NA] — Insufficient number of events to calculate using the K-M method

15. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first dose of study drug until the date of death (any reason). If the participant is alive or the vital status is unknown, the participant will be censored at the date the participant was last known to be alive.
Time Frame: From the first patient first visit to 8 months after the last patient first visit (about 48 months)
Population: All Treated Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Months | 13.31 [6.57 to 15.87] | 11.07 [5.16 to 15.31] | 37.16 [18.63 to NA] — Insufficient number of participant deaths to calculate upper limit number through the K-M Method | NA [0.07 to NA] — Insufficient number of participant deaths to calculate median and upper limit number through the K-M Method | NA [NA to NA] — Insufficient number of participant deaths to calculate median, lower limit number and upper limit number through the K-M Method

16. Post Hoc Outcome: Safety Analysis - Number of Participant Deaths - Extended Collection
Description: Number of participant Deaths
  This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 30-March-2022)
Time Frame: from first date of treatment to final database lock. Approximately 6 years and 7 months.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 30 | 26 | 14 | 4 | 8

17. Post Hoc Outcome: Safety Analysis - Number of Participants With Adverse Events - Extended Collection
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
  This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 30-March-2022)
Time Frame: From first patient first treatment to first to 100 days post last treatment. Approximately 6 years and 4 months.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 42 | 33 | 29 | 10 | 30

18. Post Hoc Outcome: Safety Analysis - Number of Participants With Serious Adverse Events - Extended Collection
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * results in death
  * is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  * requires inpatient hospitalization or causes prolongation of existing hospitalization.
  * results in persistent or significant disability/incapacity
  * is a congenital anomaly/birth defect
  * is an important medical event This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 30-March-2022)
Time Frame: From first patient first treatment to first to 100 days post last treatment. Approximately 6 years and 4 months.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 22 | 19 | 14 | 4 | 10

19. Post Hoc Outcome: Safety Analysis - Number of Participants With Adverse Events Leading to Discontinuation - Extended Collection
Description: Number of Adverse events leading to discontinuation
  This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 30-March-2022)
Time Frame: From first patient first treatment to first to 100 days post last treatment. Approximately 6 years and 4 months.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 12 | 11 | 10 | 2 | 9

20. Post Hoc Outcome: Safety Analysis - Number of Participants With Drug Related Adverse Events - Extended Collection
Description: Number of Drug Related Adverse Events
  This outcome measure represents an updated version of the primary endpoint to include additional data collection that has occurred after the primary completion date. (Assessments were made until 30-March-2022)
Time Frame: From first patient first treatment to first to 100 days post last treatment. Approximately 6 years and 4 months.
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Diffuse Large B-cell Lymphoma (DLBCL) | Peripheral T-cell Lymphoma (PTCL) | Cutaneous T-cell Lymphoma (CTCL) | Mediastinal Grey Zone Lymphoma (MGZL) | Primary Mediastinal B-cell Lymphoma (PMBL)
Number analyzed (Participants) | 42 | 33 | 29 | 10 | 30
Participants | 35 | 28 | 26 | 9 | 25

ADVERSE EVENTS:
Time Frame: From first patient first visit to first to final data base lock. Approximately 6 years and 7 months. All cause mortality is calculated from first treatment to final data base lock.. Approximately 6 years and 7 months.
Groups:
- DLBCL; PTCL; CTCL; MGZL; PMBL: 1.8mg/kg brentuximab vedotin (BV) + 240mg nivolumab
Arm/Group | DLBCL | PTCL | CTCL | MGZL | PMBL
All-Cause Mortality (participants affected / at risk) | 30/42 | 26/33 | 14/29 | 4/10 | 8/30
Serious Adverse Events (participants affected / at risk) | 23/42 | 25/33 | 18/29 | 5/10 | 12/30
Other Adverse Events (participants affected / at risk) | 42/42 | 33/33 | 28/29 | 9/10 | 28/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLBCL (N=42) | PTCL (N=33) | CTCL (N=29) | MGZL (N=10) | PMBL (N=30)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 10 | 2 | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 1 | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Clostridium test positive (Investigations) | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 9 | 4 | 1 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Dysmetria (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 2
Nephroangiosclerosis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DLBCL (N=42) | PTCL (N=33) | CTCL (N=29) | MGZL (N=10) | PMBL (N=30)
Anaemia (Blood and lymphatic system disorders) | 5 | 10 | 1 | 6 | 3
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 8 | 9 | 0 | 4 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 8 | 1 | 3 | 5
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 2 | 0 | 2 | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 4
Hypothyroidism (Endocrine disorders) | 1 | 1 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 10 | 9 | 1 | 0 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 2
Constipation (Gastrointestinal disorders) | 9 | 8 | 3 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 20 | 14 | 15 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 4 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 2 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 17 | 12 | 10 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 9 | 8 | 3 | 0 | 3
Asthenia (General disorders) | 11 | 7 | 5 | 0 | 4
Chest pain (General disorders) | 1 | 0 | 0 | 1 | 2
Chills (General disorders) | 7 | 2 | 2 | 0 | 2
Fatigue (General disorders) | 16 | 15 | 8 | 1 | 2
Gait disturbance (General disorders) | 1 | 0 | 1 | 1 | 0
Malaise (General disorders) | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 4 | 2 | 7 | 0 | 1
Pain (General disorders) | 1 | 1 | 0 | 0 | 4
Peripheral swelling (General disorders) | 3 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 13 | 12 | 14 | 2 | 7
Ear infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 0 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 2 | 1 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 5 | 1 | 1 | 2 | 1
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 1 | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 2 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 4 | 6 | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 6 | 2 | 2 | 1
Amylase increased (Investigations) | 1 | 3 | 3 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 3 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 2 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 1 | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 3 | 4 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 3 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 5 | 0 | 0 | 2
Platelet count decreased (Investigations) | 1 | 3 | 2 | 0 | 1
Weight decreased (Investigations) | 4 | 2 | 3 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 6 | 5 | 2 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 4 | 1 | 3 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 5 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 7 | 4 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 1 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 1 | 3
Dizziness (Nervous system disorders) | 3 | 3 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 3 | 1 | 0 | 1
Headache (Nervous system disorders) | 6 | 3 | 4 | 0 | 6
Neuropathy peripheral (Nervous system disorders) | 14 | 5 | 9 | 0 | 9
Paraesthesia (Nervous system disorders) | 3 | 5 | 1 | 3 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 5 | 3 | 2 | 5
Anxiety (Psychiatric disorders) | 3 | 2 | 2 | 0 | 2
Insomnia (Psychiatric disorders) | 5 | 1 | 4 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 3 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 6 | 3 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 4 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 0 | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4 | 2 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 2 | 0 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 10 | 8 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 5 | 9 | 4 | 0 | 6
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 3 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 3 | 3 | 2 | 0
Hypotension (Vascular disorders) | 9 | 4 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02581631/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT02581631/SAP_001.pdf